CLINICAL TRIAL: NCT01597284
Title: Oral Therapies in Oncology: Cognitive Function and Compliance
Status: Terminated | Type: Observational
Why Stopped: Loss of recruitment
Sponsor: Centre Francois Baclesse (Other)
Responsible Party: Sponsor
Other Study IDs: COG-OBS
Record Dates: First submitted 2012-05-10; First posted 2012-05-14 (Estimated); Last update posted 2017-02-10 (Actual); Status verified 2016-03

CONDITIONS: Oral Therapies; Cancer; Cognitive Function; Compliance
Keywords: Oral therapies; Cancer; cognitive function; compliance
MeSH Terms: conditions — Neoplasms; Patient Compliance

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The investigators propose to evaluate the compliance of oral cancer therapies, particularly the possible link between this observance and cognitive function of patients at initiation of treatment. To our knowledge, this study will be among the first conducted on the issue in France and is an innovative approach in the management of cancer patients. The inclusion of cognitive dysfunction is part of a comprehensive approach to improving the quality of life and fully meets the objectives of both plans cancer, including those of the axis "Living during and after cancer" highlighted in the Cancer Plan

ELIGIBILITY:
Inclusion Criteria:

* Age over 18 years,
* Patients treated with a first prescription of exclusive oral therapy (chemotherapy and/or targeted therapy) as part of a cancer,
* Patients who begin treatment with ZYTIGA ® (abiraterone acetate) are incluables,
* Patients with asymptomatic brain metastases are incluables,
* Lack of personality disorders and psychiatric illness scalable,
* Knowledge of spoken and written French,
* Having signed the informed consent of study participation.

Exclusion Criteria:

* Pathology psychiatric
* Refusal to participate,
* Patient unable to respond to cognitive tests, - Documented use of drugs,
* Heavy drinking, - Cancer primitive central nervous system, - Participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient treated for cancer by a first prescription of exclusive oral therapy (chemotherapy and / or targeted therapy)
Sampling Method: Probability Sample
Enrollment: 129 (Actual)
Dates: Start 2012-02; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Assess the relationship between cognitive function at baseline oral anti-cancer treatment and adherence to treatment. | 8 months

CONTACTS AND LOCATIONS:
Overall Officials: JOLY Florence, PhD, Principal Investigator — Centre François Baclesse
Locations (1):
- Centre François Baclesse, Caen, France